CLINICAL TRIAL: NCT05081258
Title: Influence of Presurgical Orthodontic Molding on the Growth of Newborns With Unilateral Cleft Lip Palate: a Prospective, Randomized, Clinical Trial
Brief Title: Influence of Presurgical Orthodontic Molding on the Growth of Newborns With Unilateral Cleft Lip Palate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Dr. Corinna Lesley Seidel, Orthodontist, Senior Physician, University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ER-pAM-NAM-UCLP-RCT
Record Dates: First submitted 2021-08-04; First posted 2021-10-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cleft Lip and Palate; Unilateral Cleft Lip
Keywords: passie Alveolar Molding; Nasoalveolar Molding; Maxillary Growth; Facial Asymmetry
MeSH Terms: conditions — Cleft Lip; Facial Asymmetry | interventions — Nasoalveolar Molding

STUDY DESIGN:
Intervention Model Description: prospective, longitudinal, randomized, clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAM treatment (Active Comparator): Study Group: newborns with UCLP will be treated with a palate plate with nasal stent (Nasoalveolar Molding = NAM)
  Interventions: Procedure: Nasoalveolar Molding
- pAM treatment (Sham Comparator): Control Group: newborns with UCLP will be treated with a palate plate without nasal stent (passive Alveolar Molding = pAM)
  Interventions: Procedure: passive Alveolar Molding

INTERVENTIONS:
Procedure: passive Alveolar Molding — A passive palate plate (passive Alveolar Molding) will be inserted within the first week after birth. The pAM appliance will be modified on regular appointments and remain until surgical lip closure (6-7 months of life). After surgical lip closure, infants will receive a nostril retainer and the treatment with the pAM appliance will continue until palate closure (10-12 months of life).
  Arms: pAM treatment
Procedure: Nasoalveolar Molding — A passive palate plate will be inserted within the first week after birth. A nasal stent will be added to the palate plate after one week (NAM appliance). The NAM appliance will be modified on regular appointments and remain until surgical lip closure (6-7 months of life). After surgical lip closure, infants will receive a nostril retainer and will be treated with a passive palate plate without nasal stent until palate closure (10-12 months of life).
  Arms: NAM treatment

SUMMARY:
Orofacial clefts are the second most common birth deformity and vary in etiology and phenotype, e.g. isolated cleft palate, cleft lip or cleft lip palate. Especially newborns with unilateral complete cleft lip and palate (UCLP) present severe facial asymmetries auch as a broad and flat ala of the nose, a deviation of the columella and the philtrum to the non cleft side. Since postnatal asymmetries can even remain after surgical lip closure in a alleviated shape, therapeutic presurgical orthodontic approaches to improve symmetrie of the nose and to achieve ideal conditions for lip surgery are essential.

Presurgical orthodontic treatment for newborns with UCLP start within the first days after birth to separate oral and nasal cavitiy, to improve breathing and feeding and to regulate growth of the maxillary segments using passive appliances (passive Alveolar Molding (pAM)). An advanced and widely spread concept is the Nasoalveolar Molding (NAM) by Grayson, which was first introduced in 1993 as a palate plate combined with a nasal stent as a non-invasive presurgical appliance to stimulate growth of the nose and use the postnatal potential to modulate the nasal cartilage. The aim of the NAM therapy is to reduce nasal width, to reduce deviation of the columella to the non cleft side and to increase nostril height. However, due to inhomogeneous study designs and results, so far only a slightly positive effect using NAM therapy could be detected and prospective, randomized clinical trials are necessary.

The aim of the study is to analyse and to compare the effects of pAM versus NAM treatment in newborns with UCLP in the first year of life. The following parameters will be analysed on defined study time points: nostril width, nasal morphology, cleft width, maxillary growth, statical and dynamical facial asymmetries and facial perception.

ELIGIBILITY:
Inclusion Criteria:

* newborns/infants with non-syndromal (ns) unilateral cleft lip palate (UCLP)
* signed informed consent by the parents or legal guardian

Exclusion Criteria:

* newborns/infants with syndromal (s) unilateral cleft lip palate (UCLP)
* insufficient adherence and compliance by the parents or legal guardian
* withdrawal of informed consent by the parents or legal guardian

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Columella Deviation Angle | From baseline (after birth) until surgical lip closure (6 - 7 months of life)
  The change of the Collumella Deviation Angle from Baseline until surgical lip closure. The change of the Columella Deviation Angle will be measured digitally using 3D-scanned models from the nose (scans and impressions from the nose) and defined anatomical points placed by four raters.
  Sbalc (lNc) = Subalar point on the cleft side Sbalnc (lNnc) = Subalar point on the non-cleft side SN = Subnasal point sn'c (mNc) = Subnasale' point Prn = Pronasal point
  CDA = Columella Deviation Angle = Angle (°) between the columella axis (connecting line between SN and Prn) and Subalar base line (connecting line between Sbalc and Sbalnc) on the cleft side
Nostril Width on the cleft side | From baseline (after birth) until surgical lip closure (6 - 7 months of life)
  The change of the Nostril Width on the cleft side from Baseline until surgical lip closure considering different time points. The change of the Nostril Width on the cleft side will be measured digitally using 3D-scanned models from the nose (scans and impressions from the nose) and defined anatomical points placed by four raters:
  Sbalc (lNc) = Subalar point on the cleft side Sbalnc (lNnc) = Subalar point on the non-cleft side SN = Subnasal point sn'c (mNc) = Subnasale' point Prn = Pronasal point NWc = Nostril Width on the cleft side = Distance (mm) of the connecting line between Sbalc and sn'c

SECONDARY OUTCOMES:
Nasal shape | From baseline (after birth) until one year after surgical palate closure (24 months of life)
  The change of the nasal shape from Baseline until one year after surgical palate closure considering different time points. The change of the nasal shape will be measured digitally using 3D-scanned models from the nose (scans and impressions from the nose) and defined anatomical points placed by four raters and used for distance (mm) measurements: Subalar point; Subnasal point; Lip Points; ala of the nose; cranial point of the nostril and medial point of the nostril.
Nasal symmetry | From baseline (after birth) until one year after surgical palate closure (24 months of life)
  The change of the nasal symmetry from Baseline until one year after surgical palate closure considering different time points. The change of the nasal symmetry will be measured digitally using 3D-scanned models from the nose (scans and impressions from the nose) and defined anatomical points placed by four raters and used for angle (°) measurements: Subalar point; Subnasal point; Lip Points; ala of the nose; cranial point of the nostril and medial point of the nostril.
Alveolar cleft width and transversal/sagittal maxillary growth | From baseline (after birth) until one year after surgical palate closure (24 months of life)
  The change of the anterior cleft width and transversal/sagittal maxillary growth from Baseline until one year after surgical palate closure considering different time points. The change of the alveolar cleft width and transversal/sagittal maxillary growth will be measured digitally using 3D-scanned models from the maxilla (impressions from the maxilla) and defined anatomical points placed by four raters and used for distance (mm) measurements:
  pole points; mesial/distal canine points; tuber points and incisal point.
Alveolar symmetry and rotation of alveolar segments | From baseline (after birth) until one year after surgical palate closure (24 months of life)
  The change of the alveolar symmetry and rotation of alveolar segments from Baseline until one year after surgical palate closure considering different time points. The change of the alveolar symmetry and rotation of alveolar segments will be measured digitally using 3D-scanned models from the maxilla (impressions from the maxilla) and defined anatomical points placed by four raters and used for angle (°) measurements:
  pole points; mesial/distal canine points; tuber points and incisal point.
Statistical and dynamical facial asymmetries | From baseline (after birth) until one year after surgical palate closure (24 months of life)
  The change of statical and dynamical facial asymmetries from Baseline until one year after surgical palate closure considering different time points. The statical and dynamical facial asymmetries will be measured digitally using 3D-scans of the face performed on 5 time points (1. rest position, 2. between 1 and 3, 3. maximal facial expression, 4. between 3 and 5, 5. final rest position). Defined anatomical an constucted points will be placed by four raters. Measurements will be performed by mirroring scans accordind to a reference plane. Asymmetries are the distances (mm) of the corresponding Points, which would be 0mm in perfect symmetry.
  The following points will be placed: S = Superciliar Point, Exocanthion; Endocanthion; Zygion; Glabella; Nasion; Pronasale; Subnasale; Pogonion; Subalare; Alare; Cheilion; Labrale superius; Labrale inferius; Crista philtri and Lip Points (median, lateral, corresponding points).
Facial perception | From Baseline (after birth) until surgical lip closure (6-7 months of life)
  Facial perception will be rated using 3 pictures photographs / processed photographs of each newborn with UCLP within the first weeks after birth, after insertion of first appliance and until surgical lip closure (without NAM appliance, with NAM appliance, without cleft processed using photoshop). The pictures will be rated from laypersons using a 10-point-rating scale ranging from 1 to 10.
  1 = highest attractiveness (greatest positive emotional valance) 10 = least attactiveness / Aversion (greatest negative emotional valence).

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Seidel, Dr., Study Director — Department of Orthodontics and Orofacial Orthopedics, University Hospital of Erlangen-Nurnberg; Lina Gölz, Prof. Dr., Study Director — Department of Orthodontics and Orofacial Orthopedics, University Hospital of Erlangen-Nurnberg; Karin Strobel, Dr., Study Director — Department of Orthodontics and Orofacial Orthopedics, University Hospital of Erlangen-Nurnberg
Locations (1):
- Department of Orthodontics and Orofacial Orthopedics, University Hospital of Erlangen-Nurnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No